CLINICAL TRIAL: NCT02967172
Title: Efficacy of Multimodal Periarticular Injections in Operatively Treated Ankle Fractures: A Randomized Controlled Trial
Brief Title: Efficacy of Multimodal Periarticular Injections in Operatively Treated Ankle Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201608737
Record Dates: First submitted 2016-10-27; First posted 2016-11-18 (Estimated); Results first posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Pain, Postoperative; Ankle Fractures
MeSH Terms: conditions — Pain, Postoperative; Ankle Fractures | interventions — Ropivacaine; Epinephrine; Morphine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Peri-incisional injection (Experimental): A single, 25 cc multimodal analgesic cocktail will be injected following completion of ankle fracture fixation/instrumentation while the patient remains under general anesthesia and prior to skin closure. The injection will be administered as such:
  * 20 mL injected into the peri-incisional soft tissues in a circumferential fashion
  * 5mL injected into the ankle joint This cocktail includes 200 mg of 0.8% ropivacaine, 0.6 mg of epinephrine, 5 mg of morphine sulfate, and sodium chloride solution. All infiltrations will be completed with a blunt trochar to minimize the risk of intravascular injection.
  Interventions:
  Drug: Ropivacaine Drug: Epinephrine Drug: Morphine Drug: 0.9% sodium chloride solution Following surgery, patients in the treatment and non-treatment groups will both be provided with the same intravenous (patient-controlled analgesia) and oral pain medications scheduled "per needed".
  Interventions: Drug: Ropivacaine; Drug: Epinephrine; Drug: Morphine; Drug: 0.9% sodium chloride solution
- Control (No Intervention): Ankle fracture fixation/instrumentation will be completed per the standard of care. No peri-incisional injection will be completed.

INTERVENTIONS:
Drug: Ropivacaine
  Other Names: Naropin
  Arms: Peri-incisional injection
Drug: Epinephrine
  Other Names: Adrenalin
  Arms: Peri-incisional injection
Drug: Morphine
  Other Names: Duramorph
  Arms: Peri-incisional injection
Drug: 0.9% sodium chloride solution
  Other Names: 0.9% normal saline
  Arms: Peri-incisional injection

SUMMARY:
The purpose of this study is to determine the efficacy and safety of a peri-articular multimodal injection for post-operative pain control following operative management of closed, rotational ankle fractures. Enrolled subjects will be randomized to either receive or not receive intra-operative injections in addition to standard opioid analgesic regimens. Patients will be treated with standard of care surgical techniques by the treating orthopaedic surgeon for the patient's specific fracture pattern. The patients randomized into the injection cohort will receive a 25cc intra-operative injection with 200 mg ropivacaine, 0.6 mg epinephrine, 5 mg and morphine into the local superficial and deep peri-incisional tissues while under general anesthesia. Total post-operative opioid consumption expressed in morphine equivalent dose will be recorded, including IV and oral opioids. Time in hours from operation conclusion to discharge and discharge disposition (to where the patient is discharged) will also be recorded. Post-operative pain scores will be assessed and recorded in the immediate post-operative period and every 4 hours subsequently until the patient is discharged. Medication related side effects will be monitored. The investigators hypothesize that the injection cohort will have reduced pain scores, lower narcotic requirements, shorter length of stay, and be more likely to discharge to home following surgery.

DETAILED DESCRIPTION:
Periarticular fractures (bone breaks extending into the joint surface) treated by orthopaedic surgeons are associated with significant pain in the post-operative period, often requiring high doses of opioid analgesics. In recent years, the high risk of misuse, abuse, and death associated with prescription opioid use has become increasingly evident.

Although physicians are being advised to avoid administration of opioid prescriptions, alternative pain management options are limited. Currently, there is a need to investigate different pain management models in order to provide safe and effective pain relief during the post-operative period. The investigators aim to evaluate the effectiveness of peri-incisional multimodal injections as an alternative post-operative pain control method in orthopaedic trauma patients with operative ankle fractures. Approximately 200 patients will be randomized to either receive or not receive intra-operative injections in addition to standard opioid analgesic regimens. Post-operative pain management outcomes will be assessed and compared between the 2 study groups to determine effectiveness of the injections. The proposed study will build upon related work to advance post-operative pain control regimens in orthopaedic surgery. Goals include the reduction of unnecessary patient suffering, reliance on opioids, and length of stay, while improving patient experience. These aims will be accomplished through the expansion of currently used multimodal periarticular injections from populations undergoing elective surgery to orthopaedic trauma patients with rotational ankle fractures.

The study design is a prospective, double-blinded, randomized controlled trial. Patients included in the study will be randomly assigned to one of two treatment groups: intra-operative multimodal periarticular injection or control (no injection). The peri-incisional injection will consist of ropivacaine, epinephrine, and morphine. All pharmacologic agents in the anesthetic cocktail are FDA approved and have been previously used in combination during other types of orthopaedic surgeries.

All patients included in the study will receive standard post-operative opioid analgesic regimens, administered 'per needed', regardless of their assigned treatment group per study protocol. ≥ 40 patients will be randomly assigned to each group. The patients enrolled in the investigation as well as health care professionals performing post-operative assessments and collecting data will be blinded to treatment allocation. The feasibility of multimodal peri-incisional injections is supported by their current efficacy in populations undergoing elective orthopedic surgeries. These injections may be equally effective at reducing pain compared to regional anesthesia with continuous infusions, and single-shot nerve blocks.

The investigators hypothesize that the injection cohort will have reduced pain scores, lower narcotic requirements, shorter length of stay, and be more likely to discharge to home following surgery.

ELIGIBILITY:
Inclusion Criteria:

* All consenting patients 18 years of age and older with operative, closed, rotational ankle fractures treated with internal fixation.

Exclusion Criteria:

* Patients with any of the following:

  * Allergy or medical contraindication to any of the study medications
  * Pregnant women
  * Diagnosed dementia
  * Preexisting opioid or illicit drug dependency
  * Major neuromuscular deficit
  * Severe systemic disorder (heart failure, respiratory failure, kidney failure, liver failure, or a clotting disorder)
  * Major head trauma
  * Concomitant distracting injury
  * Other surgical intervention in the study period (1 week)
  * Revision operations
  * Insists to receive peripheral nerve blocks for surgical anesthesia
  * Refusal to participate

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Hancock, MD, Principal Investigator — Resident Physician
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Peri-incisional Injection: * 20 mL injected into the peri-incisional soft tissues in a circumferential fashion
  * 5mL injected into the ankle joint This cocktail includes 200 mg of 0.8% ropivacaine, 0.6 mg of epinephrine, 5 mg of morphine sulfate, and 0.9% sodium chloride solution.
- Control: No peri-incisional injection will be completed during surgical fixation/instrumentation
Period: Overall Study
Arm/Group | Peri-incisional Injection | Control
Started | 49 | 51
Completed | 49 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Peri-incisional Injection: A single, 25 cc multimodal analgesic cocktail will be injected following completion of ankle fracture fixation/instrumentation while the patient remains under general anesthesia and prior to skin closure. The injection will be administered as such:
  * 20 mL injected into the peri-incisional soft tissues in a circumferential fashion
  * 5mL injected into the ankle joint This cocktail includes 200 mg of 0.8% ropivacaine, 0.6 mg of epinephrine, 5 mg of morphine sulfate, and sodium chloride solution. All infiltrations will be completed with a blunt trochar to minimize the risk of intravascular injection.
  Interventions:
  Drug: Ropivacaine Drug: Epinephrine Drug: Morphine Drug: 0.9% sodium chloride solution Following surgery, patients in the treatment and non-treatment groups will both be provided with the same intravenous (patient-controlled analgesia) and oral pain medications scheduled "per needed".
  Ropivacaine
  Epinephrine
  Morphine
  0.9% sodium chloride solution
- Total: Total of all reporting groups
Arm/Group | Peri-incisional Injection | Control | Total
Number analyzed (Participants) | 49 | 51 | 100
Age, Customized [Median (Full Range); unit: years]
  Age range | 40 [20 to 80] | 41 [18 to 80] | 40 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 19 | 21 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Age [Mean (Standard Deviation); unit: years] | 45.4 (17.6) | 43.7 (17.6) | 44.6 (17.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Post-operative Visual Analog Pain Scores (VAS)
Description: The primary outcome was VAS pain over the first 48 hours postoperatively. Patients reported pain with use of a 100-mm VAS, with 0-mm being no pain and 100-mm being the most extreme pain imaginable. A higher score indicates worse pain. Scores were reported as mean values at 24 hours post-surgery and 48 hours post-surgery.
Time Frame: Immediately following surgery, then every 4 hours following surgery for 48 hours post-surgery.
Measure: Mean (Standard Deviation); unit: 0 to 100 score on a scale
Groups:
- Peri-incisional Injection: * 20 mL injected into the peri-incisional soft tissues in a circumferential fashion
  * 5mL injected into the ankle joint This cocktail includes 200 mg of 0.8% ropivacaine, 0.6 mg of epinephrine, 5 mg of morphine sulfate, and 0.9% sodium chloride solution. .
Arm/Group | Peri-incisional Injection | Control
Number analyzed (Participants) | 49 | 51
0 to 100 score on a scale
  Mean VAS score 24hr post-op | 42 (3) | 52 (3)
  Mean VAS score 48hr post-op | 41 (3) | 50 (3)

2. Secondary Outcome: Opioid Use in First 24 Hours Post-surgery
Description: Total opioid consumption expressed in morphine equivalent dose will be recorded, including IV and oral opioids, in the first 24 hours post-surgery.
Time Frame: At 24 hours post-surgery & during the total time of inpatient stay to dischage
Measure: Median (Full Range); unit: Milligrams
Arm/Group | Peri-incisional Injection | Control
Number analyzed (Participants) | 49 | 51
Milligrams
  Opioid use 24hr post-surgery | 25.5 [0 to 74.7] | 28.3 [2.5 to 91.0]
  Total inpatient opioid use | 29.0 [0 to 85.3] | 32.7 [4.3 to 215.0]

3. Secondary Outcome: Post-operative Length of Stay
Description: Number of days in the hospital following surgery
Time Frame: From immediately following surgery to 90 days after.
Measure: Median (Full Range); unit: Hours
Arm/Group | Peri-incisional Injection | Control
Number analyzed (Participants) | 49 | 51
Hours | 22.3 [1.7 to 182.3] | 22.5 [2.2 to 123.3]

4. Secondary Outcome: Patients Returning Home Following Surgery
Description: Number of patients returning to their home following discharge, vs. going to a rehabilitation or skilled nursing facility
Time Frame: Following hospital discharge from surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Peri-incisional Injection | Control
Number analyzed (Participants) | 49 | 51
Participants | 49 | 46

5. Other Pre Specified Outcome: Medication-related Side Effects
Description: Patients will be monitored by nursing personnel for medication side effects related to ropivacaine toxicity including blurred vision, hearing problems, transient peripheral paralysis, dizziness, convulsion, uncontrolled muscle contraction, hypotension, bradycardia, and new onset arrhythmia.
Time Frame: From immediately following surgery to 7 days after.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through study completion, average 6 months
Arm/Group | Peri-incisional Injection | Control
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 0/49 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT02967172/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT02967172/SAP_001.pdf